CLINICAL TRIAL: NCT02415114
Title: An Open Label Pilot Study to Evaluate the Effectiveness of Omega Q Plus® Resveratrol at Increasing Blood Levels of CoQ10 in Healthy Subjects and Subjects on Statins
Brief Title: An Open Label Study Evaluating the Effectiveness of Omega Q Plus® Resveratrol at Increasing Blood Levels of CoQ10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Healthy Directions, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15COHH
Record Dates: First submitted 2015-03-03; First posted 2015-04-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: CoQ10 Blood Levels; CoQ10 Blood Levels With Statin Use
Keywords: Coenzyme Q10; Resveratrol; Statin
MeSH Terms: interventions — Resveratrol; coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Population (Active Comparator): Healthy Population with Omega Q Plus Resveratrol (with 50mg CoQ10)
  Interventions: Dietary Supplement: Omega Q Plus Resveratrol (with 50mg CoQ10)
- Population taking Statins (Active Comparator): Population taking Statins with Omega Q Plus Resveratrol (with 50mg CoQ10)
  Interventions: Dietary Supplement: Omega Q Plus Resveratrol (with 50mg CoQ10)

INTERVENTIONS:
Dietary Supplement: Omega Q Plus Resveratrol (with 50mg CoQ10) — Omega Q Plus Resveratrol (with 50mg CoQ10)

SUMMARY:
The primary objective of this study is to assess the blood levels of Coenzyme Q10 in healthy subjects when administered Omega Q Plus® Resveratrol for 28 days.The secondary objective of the study is to determine if statin use has an impact on the blood levels of Coenzyme Q10 when administered Omega Q Plus® Resveratrol for 28 days. The safety objectives will include assessment of safety evaluations as determined by:

* laboratory tests - CBC, electrolytes (Na, K, Cl), glucose, creatinine, AST, ALT, GGT, and bilirubin
* vital signs - heart rate and blood pressure
* adverse events

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy adults

* Male or female 45 years of age or older
* BMI <30kg/m2 (±1 kg/m2)
* If female, subject is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

OR Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include: Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System). Double-barrier method. Non-hormonal intrauterine devices. Vasectomy of partner. Non-heterosexual lifestyle (same-sex relationship).

* CoQ10 levels between 0.5 mcg/mL - 1 mcg/mL
* Agree to maintain current level of physical activity, caffeine consumption habits, alcohol consumption habits, smoking habits and dietary habits throughout the study
* Has given voluntary, written, informed consent to participate in the study

Inclusion criteria for adults on statin medications

* Adults on statin medications for at least 3 months and are otherwise healthy
* Male or female 45 years of age or older
* BMI <30kg/m2 (±1 kg/m2)
* If female, subject is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

OR Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System). Double-barrier method. Non-hormonal intrauterine devices. Vasectomy of partner.Non-heterosexual lifestyle (same-sex relationship)

* Agree to maintain current level of physical activity, caffeine consumption habits, alcohol consumption habits, smoking habits and dietary habits throughout the study
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

Exclusion criteria for healthy adults

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Unstable medical conditions
* History of atrial or ventricular arrhythmia
* History of atherosclerosis
* History of seizures
* Type I or Type II diabetes
* Use of illicit drugs or history of alcohol or drug abuse within the last 6 months
* Currently having more than 2 standard alcoholic drinks per day
* Medical use of marijuana
* Clinically significant abnormal laboratory results at screening
* History or a current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subject with cancer in full remission more than 5 years after diagnosis are acceptable
* Use of prescription blood thinner medications (i.e. warfarin etc.)
* Use of products containing CoQ10 other than vitamins or minerals within 2 weeks of randomization
* Uncontrolled hypertension defined as untreated systolic blood pressure >160 mmHg or/or diastolic blood pressure >100mmHg
* Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
* Significant abnormal liver function as defined as AST or/ALT > 2 times the upper limit of normal (ULN), and/or bilirubin > 2 times the ULN
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to study supplement ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Exclusion criteria for adults on statins

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Conditions that in the opinion of the investigator may suggest that the subject may be unsuitable for this study
* Unstable medical conditions
* Use of illicit drugs or history of alcohol or drug abuse within the last 6 months
* Currently having more than 2 standard alcoholic drinks per day
* Medical use of marijuana
* Clinically significant abnormal laboratory results at screening (except elevated levels of creatinine kinase that will be considered based on the opinion of the Investigator)
* History or a current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subject with cancer in full remission more than 5 years after diagnosis are acceptable
* History of muscle disease unrelated to statin use
* History of seizures
* Any acute disease that may influence plasma CoQ10 levels
* Subjects on background CoQ10 therapy during the last 3 months
* Use of products containing CoQ10 other than vitamins or minerals within 2 weeks of randomization
* Uncontrolled hypertension defined as untreated systolic blood pressure >160 mmHg or/or diastolic blood pressure >100mmHg
* Use of prescription blood thinner medications (i.e. warfarin etc.)
* Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
* Significant abnormal liver function as defined as AST or/ALT > 2 times the upper limit of normal (ULN), and/or bilirubin > 2 times the ULN
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to study supplement ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To assess the blood levels of Coenzyme Q10 in healthy subjects when administered Omega Q Plus® Resveratrol for 28 days. | 28 days

SECONDARY OUTCOMES:
Change from Baseline in blood levels of Coenzyme Q10 at 28 days | 28 days

OTHER OUTCOMES:
Change from,14 days prior to Baseline, in safety blood chemistry parameters (glucose, creatinine, AST, ALT, GGT, bilirubin) at 28 days | 42 days
Change from,14 days prior to Baseline, in vital signs at 28 days | 42 days
Number of Participants with Adverse Events | 42 days
Change from,14 days prior to Baseline, in hematology parameters (CBC, electrolytes) to 28 days | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada